CLINICAL TRIAL: NCT05688059
Title: Is Absorbable Suture Non-Inferior to Permanent Suture in Sacrospinous Ligament Suspension? A Randomized Controlled Trial
Brief Title: Absorbable Suture vs Permanent Suture in Sacrospinous Ligament Suspension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Laura Dhariwal, MD, Principal Investigator, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1963079-1
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Organ Prolapse; Uterovaginal Prolapse; Vaginal Vault Prolapse; Cystocele
Keywords: Sacrospinous Ligament Suspension; Permanent Suture; Absorbable Suture; Efficacy; Suture-related Complications
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Absorbable Suture (Experimental): Absorbable suture for sacrospinous ligament suspension
  Interventions: Other: Absorbable Suture and Permanent Suture
- Permanent Suture (Experimental): Permanent suture for sacrospinous ligament suspension
  Interventions: Other: Absorbable Suture and Permanent Suture

INTERVENTIONS:
Other: Absorbable Suture and Permanent Suture — Absorbable Suture and Permanent Suture

SUMMARY:
Sacrospinous ligament suspension (SSLS) was first described in 1958. It is commonly performed for correction of apical prolapse. A combination of delayed absorbable and/or permanent sutures are commonly used for the procedure. When permanent sutures are used, risk of suture-related complications is present and patients may require suture removal. In available literature, there is limited data comparing the efficacy and suture-related complications when using different types of sutures. A previous randomized controlled trial demonstrated that using an absorbable suture is equally efficacious as delayed absorbable sutures in SSLS. However, there is no comparison to absorbable versus permanent suture. Our aim is to compare the absorbable suture versus permanent suture for treating pelvic organ prolapse and to compare suture-related complications.

Our primary outcome is comparing POPQ point C at 12 month follow up for absorbable vs permanent suture.

Participants will be randomized 1:1 to absorbable or permanent suture. Follow up will occur at 2-4 weeks, 12 weeks and 12 months after the surgery.

DETAILED DESCRIPTION:
Patient demographics, previous medical and surgical history, baseline physical exam including POP-Q will be collected from the electronic medical record following enrollment. This information will be stored in REDCap which is a secure database system.

Patients will be randomized by in REDCap system with the sequence of 1:1 with blocks of 6.

Patients and assessors will be blinded to the type of suture that was used. The surgeons will not be blinded.

All procedures will be performed by a fellowship-trained, Female Pelvic Medicine and Reconstructive Surgery board-certified surgeon.

Sacrospinous ligament suspension (SSLS) procedure with the assigned suture and any scheduled concomitant prolapse and anti-incontinence procedures will be performed.

Follow up exams will occur at 2-4 weeks, 12 weeks and 12 months post-operatively. The follow up visits will include a POP-Q exam at 12 weeks and 12 months. The 12 months follow up visit will include a PGI-I questionnaire. All participants will also be assessed for any suture-related complications. 12 month POP-Q exam will be completed by one of the providers who will be blinded to the suture type.

There will be no additional follow up visits for participation in the study. The follow up appointments at 2-4 weeks, 12 weeks and 12 months are the times of usually scheduled post-operative follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Females
* Patients of Atlantic Urogynecology Associates undergoing sacrospinous ligament suspension procedure at Morristown and Overlook Medical Centers

Exclusion Criteria:

* Patients who did not undergo sacrospinous ligament suspension procedure based on surgeon's intraoperative decision
* Patients with current gynecologic malignancies
* Patients with history of pelvic radiation
* Patients with history of prolapse repair surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) exam Point C | 12 months
  Point C represents either the most distal edge of the cervix or the leading edge of the vaginal cuff after total hysterectomy. A provider who is blinded to the type of suture used will conduct postop POPQ exam.

SECONDARY OUTCOMES:
Prolapse Recurrence | 12 months
  Defined as: Prolapse symptoms reported by patient, Prolapse beyond the hymen on examination in any compartment , Apical prolapse ≥ ½ TVL, Reoperation or pessary use for prolapse during the study period
PGI-I | 12 months
  patient's global impression of symptom improvement
Suture-related Complications | 12 months
  presence of abnormal vaginal discharge, vaginal spotting, post-coital spotting, dyspareunia, if they can feel sutures. On the physical exam, patients will be evaluated for apical granulation tissue, and apical suture exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dhariwal, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber MD, Maher C. Epidemiology and outcome assessment of pelvic organ prolapse. Int Urogynecol J. 2013 Nov;24(11):1783-90. doi: 10.1007/s00192-013-2169-9. PMID 24142054
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Beer M, Kuhn A. Surgical techniques for vault prolapse: a review of the literature. Eur J Obstet Gynecol Reprod Biol. 2005 Apr 1;119(2):144-55. doi: 10.1016/j.ejogrb.2004.06.042. PMID 15808370
- [Background] Tseng LH, Chen I, Chang SD, Lee CL. Modern role of sacrospinous ligament fixation for pelvic organ prolapse surgery--a systemic review. Taiwan J Obstet Gynecol. 2013 Sep;52(3):311-7. doi: 10.1016/j.tjog.2012.11.002. PMID 24075365
- [Background] Jelovsek JE, Barber MD, Brubaker L, Norton P, Gantz M, Richter HE, Weidner A, Menefee S, Schaffer J, Pugh N, Meikle S; NICHD Pelvic Floor Disorders Network. Effect of Uterosacral Ligament Suspension vs Sacrospinous Ligament Fixation With or Without Perioperative Behavioral Therapy for Pelvic Organ Vaginal Prolapse on Surgical Outcomes and Prolapse Symptoms at 5 Years in the OPTIMAL Randomized Clinical Trial. JAMA. 2018 Apr 17;319(15):1554-1565. doi: 10.1001/jama.2018.2827. PMID 29677302
- [Background] Hamdy MA, Ahmed WAS, Taha OT, Abolill ZM, Elshahat AM, Aboelroose AA. Late suture site complications of sacrospinous ligament fixation. Eur J Obstet Gynecol Reprod Biol. 2019 Nov;242:126-130. doi: 10.1016/j.ejogrb.2019.08.024. Epub 2019 Sep 19. PMID 31585239
- [Background] Sailesh Ray, Atin Halder, Mimi Gangopadhyay, Saswati Halder, and Partha Pratim Pal.Comparison of Two Different Suture Materials for Transvaginal Sacrospinous Fixation of the Vault: A Prospective Randomized Trial. Journal of Gynecologic Surgery.Dec 2013.281-286.http://doi.org/10.1089/gyn.2012.0150
- [Background] Kowalski JT, Genadry R, Ten Eyck P, Bradley CS. A randomized controlled trial of permanent vs absorbable suture for uterosacral ligament suspension. Int Urogynecol J. 2021 Apr;32(4):785-790. doi: 10.1007/s00192-020-04244-1. Epub 2020 Feb 11. PMID 32047968
- [Background] Luck AM, Galvin SL, Theofrastous JP. Suture erosion and wound dehiscence with permanent versus absorbable suture in reconstructive posterior vaginal surgery. Am J Obstet Gynecol. 2005 May;192(5):1626-9. doi: 10.1016/j.ajog.2004.11.029. PMID 15902168
- [Background] Barber MD, Brubaker L, Burgio KL, Richter HE, Nygaard I, Weidner AC, Menefee SA, Lukacz ES, Norton P, Schaffer J, Nguyen JN, Borello-France D, Goode PS, Jakus-Waldman S, Spino C, Warren LK, Gantz MG, Meikle SF; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Comparison of 2 transvaginal surgical approaches and perioperative behavioral therapy for apical vaginal prolapse: the OPTIMAL randomized trial. JAMA. 2014 Mar 12;311(10):1023-34. doi: 10.1001/jama.2014.1719. PMID 24618964